CLINICAL TRIAL: NCT00006198
Title: Chronic Thalidomide Administration in Patients Undergoing Chemoembolization for Unresectable Hepatocellular Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: NCRR-M01RR00096-0958; M01RR000096 (NIH)
Record Dates: First submitted 2000-09-09; First posted 2000-09-11 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-01

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Thalidomide; Doxorubicin; Collagen

INTERVENTIONS:
Drug: thalidomide
Procedure: chemoembolization with doxorubicin/collagen

SUMMARY:
This is a clinical trial to test the safety and efficacy of the drug thalidomide in combination with a procedure called chemoembolization in patients with inoperable liver cancer. Chemoembolization is the process by which chemotherapy is instilled directly into the blood vessels feeding the tumor, so that the blood vessels feeding the tumor may be blocked. Chemoembolization consists of two separate procedures. It will be done by infusing chemotherapy with the drug doxorubicin through the hepatic artery into the liver and then by infusing collagen to cut off the blood supply to the tumor. A catheter will be inserted at various times to allow for these infusions.

The objectives are to investigate the feasibility and potential activity of chronic administration of thalidomide in patients with unresectable hepatocellular cancer who receive chemoembolization to predominant tumor masses. The toxicity of thalidomide in these patients will be evaluated. Overall safety will also be assessed. Serum levels of angiogenic cytokines such as VEGF, bFGF, and TNF-a, that are believed to have a role in hepatocellular carcinoma, will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable hepatocellular carcinoma.
* MRI of liver must show discrete tumor nodules. Lesions on angiography must be hypervascular.
* Patient must have the following minimum labs: ANC> 1200/mm3; Hemoglobin > 8 mg/dl; platelets > 50,000 mm3; hepatic transaminases < 5x normal; bilirubin < 3.0 mg/dl; and creatinine < 1.5 mg/dl.
* ECOG performance status > 2.
* No history of prior chemotherapy or biologic therapy for hepatocellular carcinoma.
* No other history of malignancy other than curatively resected basal cell carcinoma of the skin or carcinoma in situ of the cervix.
* Patients must not be pregnant or lactating.
* Sexually active men and women of childbearing age must use adequate contraception. All patients must understand the potential for severe birth defects with thalidomide and must be able to follow instructions to avoid conception while taking thalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Kaplan Comprehensive Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Wu J, Ng J, Christos PJ, Goldenberg AS, Sparano J, Sung MW, Hochster HS, Muggia FM. Chronic thalidomide and chemoembolization for hepatocellular carcinoma. Oncologist. 2014 Dec;19(12):1229-30. doi: 10.1634/theoncologist.2014-0283. Epub 2014 Oct 31. PMID 25361625